CLINICAL TRIAL: NCT00974051
Title: The Effect of Using Terbutaline or a Reduction in Basal Insulin Infusion as a Therapeutic Agent to Prevent Delayed Nocturnal Hypoglycemia in Children and Adolescents With Type 1 Diabetes
Brief Title: Use of Terbutaline or a Reduction in Basal Insulin in the Prevention of Nocturnal Hypoglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 07-0392
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-08

CONDITIONS: Type 1 Diabetes
Keywords: Children; Exercise; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Terbutaline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Subjects complete the same exercise routine, however no treatment is given at 9:00pm.
  Interventions: Other: Control
- Terbutaline (Experimental): Subjects complete same exercise routine. At 9:00pm, an oral dose of 2.5 mg of Terbutaline is administered.
  Interventions: Drug: Terbutaline
- 20% Basal Insulin Reduction (Experimental): All subjects complete the same exercise session. At 9:00pm, subject's basal rate is decreased by 20% for six hours.
  Interventions: Other: 20% basal insulin reduction

INTERVENTIONS:
Drug: Terbutaline — Oral (2.5mg) one time administration at 9:00pm
  Other Names: β2-adrenergic agonist
  Arms: Terbutaline
Other: 20% basal insulin reduction — Basal insulin rate is reduced by 20% the normal (home dose) for six hours.
  Other Names: 80% basal insulin
  Arms: 20% Basal Insulin Reduction
Other: Control — No treatment is given for the study. This arm is for comparison with the two intervention arms.
  Other Names: No intervention
  Arms: Control

SUMMARY:
The investigators hypothesize that the use of an oral dose of Terbutaline or a 20% basal reduction will be able to prevent nocturnal hypoglycemia after an afternoon exercise session. This is a randomized three period cross-over study including treatment with Terbutaline, a 20% basal reduction for six hours, or no treatment (control).

DETAILED DESCRIPTION:
In this study, a minimum of 16 youth with type 1 diabetes will be recruited. All subjects must have been diagnosed with type 1 diabetes for at least one year and on an insulin pump for at least one month. Subjects are between the ages of 10 and 17 years, inclusive, have an HbA1c less than 10.0% and normal thyroid function. Subjects can not have had a severe hypoglycemic episode in the last three months, any other illness or treatment that may affect the wearing of a continuous glucose monitor or the completion of the study as determined by the investigator. Subjects may not use drugs containing pseudoephedrine within 48 hours of the study visits.

This study consists of three overnight visits at the Clinical Translational Research Center. Meals eaten during the study will be consistent for each of the three visits.

Subjects will participate in a standardized afternoon exercise session on a treadmill as has been done in previous Diabetes Research in Children Network studies. Exercise will begin at 4pm and must be completed by 6pm. Dinner will be eaten at the end of the exercise.

At 9pm, treatment will be given as determined by the randomization group the subject is assigned to. The treatment includes either an oral dose of 2.5mg Terbutaline, a 20% basal reduction for six hours or no treatment as the control. Blood glucose levels will be measured every 30 minutes until 6am.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 1 Diabetes and using daily insulin therapy for at least one year.
* Age 10 to 17 years, inclusive.
* HbA1c < 10.0%.
* BMI 5-95th % for age and gender.
* Stable Continuous Subcutaneous Insulin Infusion regimen for at least 1 month and not anticipating a change prior to the subject's completion of the study.
* Subject uses a downloadable insulin pump.
* Normal thyroid function (measured within the previous year).
* For females, subject not intending to become pregnant during the study.
* No expectation that subject will be moving out of the area for the duration of the study.
* Informed consent form signed and understood by the parent/guardian and Child Assent form signed/understood by subjects.

Exclusion Criteria:

* The presence of a significant medical disorder (including epilepsy, or any cause of seizures other than hypoglycemia) that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol.
* A recent injury to body or limb, Addison's disease, muscular disorder or disease in the judgment of the investigator that will affect the completion of the exercise protocol.
* Asthma which has been medically treated within the last year.
* Medically diagnosed cardiac disease, hypertension, or autonomic dysfunction.
* Use of pseudoephedrine 48 hours prior to the visit (if used in the 48 hours prior to the scheduled visit, the visit will be deferred)
* Severe hypoglycemia resulting in seizure of loss of consciousness in the 3 months prior to a visit.
* Active infection (if at the time of the scheduled visit and infection is present, the visit will be deferred).
* Anticipating a significant change in exercise regimen between visits (i.e. starting or stopping an organized sport).
* Treatment with systemic or inhaled corticosteroids in the last 6 months.
* Current treatment with B-blockers or presenting with high blood pressure.
* Inpatient psychiatric treatment in the past 6 months for either the subject or the subject's primary care giver.
* Current use of oral/inhaled glucocorticoids or other medications, which in the judgment of the investigator would be a contraindication to participation in the study
* Known allergy to Terbutaline
* Treatment with atenolol (Tenormin), carteolol (Cartrol), labetalol (Normodyne, Trandate), metoprolol (Lopressor), nadolol (Corgard), phenelzine (Nardil), propranolol (Inderal), sotalol (Betapace), theophylline (Theo-Dur), timolol (Blocadren), tranylcypromine (Parnate), other medications for asthma, heart disease or depression.
* Treatment with ephedrine, phenylephrine, phenylpropanolamine, or pseudoephedrine.
* The presence of an irregular heart beat, increased heart rate glaucoma or an overactive thyroid gland.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosanna Fiallo-Scharer, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center, Aurora, Colorado, United States

REFERENCES:
- [Derived] Taplin CE, Cobry E, Messer L, McFann K, Chase HP, Fiallo-Scharer R. Preventing post-exercise nocturnal hypoglycemia in children with type 1 diabetes. J Pediatr. 2010 Nov;157(5):784-8.e1. doi: 10.1016/j.jpeds.2010.06.004. Epub 2010 Jul 21. PMID 20650471

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from the Barbara Davis Center pediatric population
Pre-assignment Details: no notes
Groups:
- Control First, Then Terbutaline, Then 20% Basal Reduction; Terbutaline First, Then 20% Basal Reduction, Then Control; 20% Basal Reduction First, Then Control, Then Terbutaline: Subjects complete the same exercise routine. No treatment is given during the Control night, Terbutaline is given at 9pm during the Terbutaline night, a 20% basal reduction is done starting at 9pm for six hours on the 20% basal reduction night.
Period: Overall Study
Arm/Group | Control First, Then Terbutaline, Then 20% Basal Reduction | Terbutaline First, Then 20% Basal Reduction, Then Control | 20% Basal Reduction First, Then Control, Then Terbutaline
Started | 6 | 4 | 6
Completed | 6 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Subjects: Subjects complete the same exercise routine. Subjects serve as there own control and participate in all interventions. No treatment is given during the Control night, Terbutaline is given at 9pm during the Terbutaline night, a 20% basal reduction is done starting at 9pm for six hours on the 20% basal reduction night.
Arm/Group | All Study Subjects
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 13.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Secondary Outcome: Percent of Nighttime Glucose Levels <80
Time Frame: 9:00pm to 6:00am
Measure: Number; unit: percentage of overnight glucose levels
Groups:
- Control Arm: No treatment is given during the Control night. Glucose levels from 9 pm to 6 am are analyzed.
- Terbutaline Arm: 2.5 mg oral terbutaline is given at 9pm during the Terbutaline night. Glucose levels from 9 pm to 6 am are analyzed.
- 20% Basal Reduction Arm: Subjects complete the same exercise routine. A 20% basal reduction is done starting at 9pm for six hours on the 20% basal reduction night. Glucose levels from 9 pm to 6 am are analyzed.
Arm/Group | Control Arm | Terbutaline Arm | 20% Basal Reduction Arm
Number analyzed (Participants) | 16 | 16 | 16
percentage of overnight glucose levels | 6.6 | 0 | 4.9

2. Secondary Outcome: Percent of Nighttime Glucose Levels <70
Time Frame: 10:00pm to 6:00am
Measure: Number; unit: percentage of nighttime glucose values
Arm/Group | Control Arm | Terbutaline Arm | 20% Basal Reduction Arm
Number analyzed (Participants) | 16 | 16 | 16
percentage of nighttime glucose values | 1.7 | 0 | 0.3

3. Secondary Outcome: Percent of Nighttime Glucose Levels >250 mg/dl
Time Frame: 10:00pm to 6:00am
Measure: Number; unit: percentage of overnght glucose values
Arm/Group | Control Arm | Terbutaline Arm | 20% Basal Reduction Arm
Number analyzed (Participants) | 16 | 16 | 16
percentage of overnght glucose values | 30.2 | 63.5 | 41.7

4. Primary Outcome: Blood Glucose Nadir
Description: BG nadir overnight after intervention
Time Frame: overnight hours
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Control Arm | Terbutaline Arm | 20% Basal Reduction Arm
Number analyzed (Participants) | 16 | 16 | 16
mg/dl | 128 (58) | 189 (60) | 162 (65)

ADVERSE EVENTS:
Groups:
- Control Arm: during control intervention night
- Terbutaline Arm: During turbutaline intervention night
- 20% Basal Reduction Arm: During 20% basal reduction night
Arm/Group | All Study Subjects | Control Arm | Terbutaline Arm | 20% Basal Reduction Arm
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes